CLINICAL TRIAL: NCT06960629
Title: The Effect of Topical Rho-kinase (ROCK) Inhibitors on Corneas of Patients With Glaucoma and Pseudophakic Bullous Keratopathy
Brief Title: The Effect of ROCK Inhibitors on Corneas of Patients With Glaucoma and Pseudophakic Bullous Keratopathy (PBK)
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Anđela Jukic, MD, PhD, University Hospital Dubrava
Other Study IDs: 2025/0327-4
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Pseudophakic Bullous Keratopathy; Glaucoma
Keywords: Glaucoma; Topical ROCK inhibitors; Netarsudil/latanoprost; corneal edema; pseudophakic bullous keratopathy (PBK)
MeSH Terms: conditions — Glaucoma; Corneal Edema | interventions — netarsudil; Latanoprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Rock inhibitor group: Group 1 or ROCK inhibitor group will receive topical netarsudil/latanoprost 1x daily for 3 months.
  Interventions: Drug: Netarsudil 0.02%/latanoprost 0.005% fixed dose combination ophthalmic solution
- Placebo group: Placebo group will receive topical placebo (artificial tear substitute) 1x daily for 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Netarsudil 0.02%/latanoprost 0.005% fixed dose combination ophthalmic solution — Patients with pseudophakic bullous keratopthy and glaucoma will receive topical netarsudil/latanoprost 1x daily for 3 months.
  Groups: Rock inhibitor group
Drug: Placebo — Patients with pseudophakic bullous keratopathy and glaucoma will receive topical placebo 8artificial tear substitute) 1x daily for 3 months.
  Groups: Placebo group

SUMMARY:
The goal of this clinical trial is to learn if topical netarsudil/latanoprost works to treat pseudophakic bullous keratopathy in patients with glaucoma. The main questions it aims to answer are:

Does topical netarsudil/latanoprost improves visual function in patients with glaucoma and pseudophakic bullous keratopathy? Does topical netarsudil/latanoprost affects the central corneal thickness (CCT) in patients with glaucoma and pseudophakic bullous keratopathy? Researchers will compare topical netarsudil/latanoprost to a placebo (a look-alike substance that contains no drug) to see if topical netarsudil/latanoprost works to treat pseudophakic bullous keratopathy (PBK).

Participants will take topical netarsudil/latanoprost or a placebo every day for 3 months and visit the clinic once every two weeks for checkups and tests.

DETAILED DESCRIPTION:
Patients with glaucoma and pseudophakic bullous keratopathy will be randomly divided in two groups. Group 1 will take topical netarsudil/latanoprost 1x daily for 3 months and group 2 will take topical placebo (artificial tear substitute) 1x daily for 3 months. Visual acuity (VA) will be evaluated using Snellen chart and converted to logarithm of the minimum angle of resolution (LogMAR). Central corneal thickness (CCT) measurements will be performed using ultrasound pacymetry (Micro Medical devices, Inc, CA). Information about adverse effects will be recorded during the study. Patients will visit every two weeks for checkups and measurements for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* both sex,
* age between 40 and 90 years
* pseudophakic bullous keratopathy
* glaucoma

Exclusion Criteria:

* other anterior segment pathology (corneal opacities);
* ocular surface inflammation
* retinal diseases affecting visual acuity

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both sex, age between 40 and 90 years with glaucoma and pseudophakic bullous keratopathy.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Visual acuity (VA) | 3 months
  Visual acuity measurements using Snellen chart and converted to logMAR

SECONDARY OUTCOMES:
Central corneal thickness (CCT) | 3 months
  CCT will be measured using ultrasound pachymetry.

CONTACTS AND LOCATIONS:
Overall Officials: Josip Pavan, MD, PhD, Study Director — University Hospital Dubrava
Locations (1):
- University Hospital Dubrava, Zagreb, Croatia, Croatia

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data.